CLINICAL TRIAL: NCT05260307
Title: Improving Spatial Perception and Speech Understanding in Multitalker Mixtures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4218E; R01DC015760 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-03-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss
Keywords: Hearing Aids; Speech Intelligibility; Spatial Hearing; Cocktail Party; Audibility; Sound Image Externalization; Speech Envelope
MeSH Terms: conditions — Hearing Loss; Speech Intelligibility

STUDY DESIGN:
Intervention Model Description: All participants will be tested under a number of experimental conditions that simulate different hearing aid conditions. They will act as their own control.
Masking Description: While participants will not be informed about the specific experimental condition being tested, certain acoustical changes may be perceptible to them and thus strict masking is impossible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental condition (Other): Participants will be presented with sound stimuli under a number of experimental conditions that simulate different hearing-aid conditions.
  Interventions: Other: hearing aid condition

INTERVENTIONS:
Other: hearing aid condition — The intervention will be a hearing aid or a modification to the sound stimulus that simulates a hearing aid configuration, style, or processing strategy.

SUMMARY:
The purpose of this study is to investigate several approaches for improving spatial perception and speech intelligibility in multitalker listening situations for hearing-aid users. The hypotheses are that spatial perception and speech intelligibility will be improved by (1) increased high-frequency audibility, (2) speech envelope enhancement, and/or (3) appropriate sound image externalization.

DETAILED DESCRIPTION:
The purpose of this study is to investigate several approaches for improving spatial perception and speech intelligibility in multitalker listening situations for hearing-aid users. Aim 1 will investigate how well different amplification strategies provide access to the spectrotemporally sparse speech information that is available in multitalker mixtures. The hypothesis is that subtle differences in high-frequency audibility across different strategies may have much greater effects on the intelligibility of sparse speech than intact speech. This Aim will involve 40 subjects with hearing loss across 2 experiments. Aim 2 is an exploratory aim that will investigate the potential of a speech enhancement algorithm to improve spatial hearing in multitalker mixtures. The hypothesis is that speech enhancement, in addition to its established monaural benefits, will enhance the salience of interaural time differences and thus provide binaural benefits in multitalker mixtures. This Aim will involve 30 subjects with normal hearing and 60 subjects with hearing loss across 3 experiments. Aim 3 will investigate how different hearing-aid styles affect sound externalization. The hypothesis is that hearing aids can disrupt sound externalization, which in turn impacts speech intelligibility in multitalker mixtures. This Aim will involve 30 subjects with normal hearing and 60 subjects with hearing loss across 3 experiments.

This is a prospective design involving adult human subjects. While the investigators will recruit subjects with normal and impaired hearing, all subjects will be assigned to the same set of experimental conditions. Therefore, for the purposes of intervention (or prospective assignment), the subjects can be treated as a single group completing the same intervention (or set of interventions). The behavioral experiments involve listening to speech sounds (either unaided, with hearing aids, or with simulated hearing aids), and providing responses related to spatial perception or speech intelligibility. The order of experimental conditions will be randomized for each subject in order to control for order effects. All of the experimental tasks and outcome measures have been previously established, have good reliability and validity, and will be appropriate for informing future studies.

ELIGIBILITY:
Inclusion Criteria: Normal-Hearing Subjects

* 18 to 35 years of age
* Audiometric thresholds that do not exceed 20 dB HL at any frequency from 250 to 8000 Hz
* Able to provide informed consent and understand experimental instructions
* Normal or corrected-to-normal vision

Inclusion Criteria: Hearing-Impaired Subjects

* 18 to 80 years of age
* Documented sensorineural hearing loss
* Able to provide informed consent and understand experimental instructions
* Normal or corrected-to-normal vision

Exclusion Criteria (some experiments)

* Non-native speakers of English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Speech intelligibility at baseline | Baseline
  Speech intelligibility scores will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in percent correct (0-100%).
Speech intelligibility post-intervention | Up to 4 hours
  Speech intelligibility scores will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in percent correct (0-100%).
Speech reception threshold at baseline | Baseline
  Speech reception thresholds will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in decibels (the level of the target speech relative to the masker speech needed to identify 50% of the words in a sentence).
Speech reception threshold post-intervention | Up to 4 hours
  Speech reception thresholds will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in decibels (the level of the target speech relative to the masker speech needed to identify 50% of the words in a sentence).
Interaural time difference discrimination at baseline | Baseline
  Thresholds for the discrimination of interaural time differences in speech will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in microseconds.
Interaural time difference discrimination post-intervention | Up to 4 hours
  Thresholds for the discrimination of interaural time differences in speech will be measured in a baseline condition (e.g. unaided) and in a number of hearing-aid conditions (post-intervention). Scale is in microseconds.
Externalization rating at baseline | Baseline
  Externalization judgments for speech will be measured in a baseline condition (e.g. unaided) and in a number of different hearing-aid conditions (post-intervention). Scale is in percent (0-100%).
Externalization rating post-intervention | Up to 4 hours
  Externalization judgments for speech will be measured in a baseline condition (e.g. unaided) and in a number of different hearing-aid conditions (post-intervention). Scale is in percent (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A Best, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in a publication will be made publicly available.
Time Frame: The data will be made available at the time of the relevant publication.